CLINICAL TRIAL: NCT02895048
Title: Clinical Effects of Cardiac Contractility Modulation (CCM) With the OPTIMIZER III System in Subjects With Heart Failure Caused by Left Ventricular Dysfunction
Brief Title: Effects of CCM-therapy in Patients With Heart Failure
Acronym: CCM-HF
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Collaborators: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Other Study IDs: ID CP OPT2009-007
Record Dates: First submitted 2011-10-07; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic heart failure
- CCM treatment: Subjects with heart failure receiving OPTIMIZER system implant

SUMMARY:
The effects of Cardiac Contractility Modulation (CCM) treatment are observed in patients with heart failure.

DETAILED DESCRIPTION:
The OPTIMIZER III System is indicated for use in patients greater than 18 years of age with symptomatic heart failure due to left ventricular systolic dysfunction despite appropriate medical therapy. The study will gather additional data on the effect of CCM treatment with the objective of determining the impact of CCM on the composite of heart failure hospitalizations and mortality in the low ejection fraction (EF < 35%) and mildly reduced ejection fraction (35 ≤ EF ≤ 45) heart failure population. The study will also assess the impact of CCM on exercise tolerance (six minute hall walk test, 6 Minute Walk Test) and quality of life (Minnesota Living With Heart Failure Questionnaire, MLWHFQ) in these same populations.

ELIGIBILITY:
Inclusion Criteria (treatment group):

* Any subject who receives an OPTIMIZER system implant and provides informed consent

Exclusion Criteria (treatment group):

* None

Inclusion Criteria (control group):

* Symptomatic heart failure (NYHA Class 2, 3 or 4) despite receiving optimal medical therapy with doses of medications that are stable (no more than 50 % variation) for at least 7 days.
* EF ≤ 45%
* Signed informed consent

Exclusion Criteria (control group):

* Heart failure due to a potentially correctible cause ( e. g. valvular disease, congenital disease)
* Idiopathic hypertrophic cardiomyopathy, restrictive or constrictive cardiomyopathy, or heart failure on the basis of a known inflammatory or infiltrative disease (e. g. amyloidosis, sarcoidosis) or constrictive disease
* Active ischemia or exercise tolerance limited by angina
* Hospitalizations for heart failure which required the use of inotropic support within 14 days of enrollment
* Chronic (permanent or persistent) atrial fibrillation or atrial flutter
* Scheduled for a CABG or a PCI procedure, or has undergone a CABG procedure within 90 days or a PCI procedure within 30 days of enrollment
* Myocardial infarction within 90 days of enrollment
* Hemodialysis or peritoneal dialysis
* Prior heart transplant
* Participating in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study shall include up to 300 subjects with CCM treatment and up to 300 subjects without CCM treatment. Patients without CCM treatment serve as Control patients and they will be recruited from centers not implanting OPTIMIZER systems.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
All-cause and cardiac mortality | 24 Months

SECONDARY OUTCOMES:
the rate of all-cause and cardiac-related hospitalizations | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Remppis, Professor, Principal Investigator — Bad Bevensen
Locations (1):
- CCB, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No